CLINICAL TRIAL: NCT02411084
Title: Prospective, Phase II/III, Randomized Clinical Study to Compare BEGEDINA® Versus "Conventional Treatment" for Treating Steroid Resistant Acute Graft-versus Host Disease
Brief Title: Study of BEGEDINA® vs "Conventional Treatment" for Treating Steroid-Resistant Acute GvHD
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Insufficient rate of accrual
Sponsor: Adienne SA (Industry)
Collaborators: ADIENNE S.r.l. S.U. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ADN011; 2015-001360-19 (EudraCT Number)
Record Dates: First submitted 2015-03-24; First posted 2015-04-08 (Estimated); Results first posted 2020-01-30 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Graft vs Host Disease
Keywords: Graft vs Host Disease; Immune System Diseases; Dipeptidyl Peptidase 4; CD4-Positive T-Lymphocytes; Hematopoietic Stem Cell Transplantation
MeSH Terms: conditions — Graft vs Host Disease; Immune System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BEGEDINA® (Begelomab) (Experimental): BEGEDINA® (Begelomab) (murine monoclonal antibody against CD26). Dose is 2.7 mg/m2/day i.v. infusion for 5 consecutive days (Study Days 1, 2, 3, 4, 5) and then single dose on each of Study Days 10, 14, 17, 21, 24 and 28, for a total of 11 doses. BEGEDINA® is supplied as 1 mg/mL concentrate for solution for infusion in vials of 6 mL (5.4 mg of active substance) for reconstitution. The total volume to be administered should be further diluted in 100 mL of 0.9% sodium chloride solution for injection prior to administration. The infusion lasts 60 minutes. Subjects are eligible for a single treatment for flare after study Day 28
  Interventions: Biological: Begelomab
- Conventional Second-line Treatment (Active Comparator): Subjects in the conventional treatment arm will receive a second line treatment, which is to be chosen by each center, based on the clinical conditions of the individual subject and according to the standard practice at the study center. Currently no treatments for this life-threatening disease have been approved in either the USA or Europe. The recommendations of the American Society for Blood and Marrow Transplantation (ASBMT) confirm that no treatment for acute steroid-refractory GvHD can be considered gold standard in terms of TRM or survival as results remain unsatisfactory and this approach has been agreed by the FDA and the EMA.
  Interventions: Biological: Conventional Second-line Treatment

INTERVENTIONS:
Biological: Begelomab — BEGEDINA® (Begelomab) is a murine immunoglobulin G (IgG) 2b monoclonal antibody against CD26 (dipeptidyl peptidase-4; DPP4) and is produced by biotechnological means.
  Other Names: BEGEDINA®
  Arms: BEGEDINA® (Begelomab)
Biological: Conventional Second-line Treatment — There are no approved second-line treatments for aGvHD and due to the life-threatening nature of the disease it was agreed with the FDA and EMA that BEGEDINA® would be compared with "best conventional second-line treatments" which will be chosen by each center, based on the clinical conditions of the individual subject and according to the standard practice at the study center and which may vary between centers. Treatments are generally biological products and could include anti-thymocyte globulin, monoclonal antibodies, such as anti-CD147, basiliximab, daclizumab and alemtuzumab; mycophenolate mofetil; anti-TNF-alpha; pentostatin; dinileukin diftitox; N-acetyl-cysteine; sirolimus; and visulizumab.
  Arms: Conventional Second-line Treatment

SUMMARY:
The objectives of this study are to determine the efficacy and safety of BEGEDINA® in subjects with steroid resistant acute graft versus host disease (GvHD). GvHD is a rare and complex immunological disease occurring in some recipients of allogeneic hematopoietic stem cell transplants (HSCTs) and affecting principally the skin, liver and gastrointestinal (GI) tissues. The disease is life threatening and may be acute or chronic and the first choice treatment for patients with acute GvHD (Grade II or higher) is the immunosuppressive corticosteroid hormone methylprednisolone. However, some GvHD patients may be resistant to this treatment leading to disease progression and a high rate of morbidity and mortality, primarily from infections and/or multi-organ failure. There are currently no other satisfactory therapies. BEGEDINA® is a therapeutic monoclonal antibody that recognises and binds to CD26 on CD4+ T lymphocytes. BEGEDINA® reduces the activity of CD26 in these cells and inhibits the immune response leading to improvement in patients that have shown steroid resistance. This study is therefore aimed at demonstrating that BEGEDINA® is a safe and effective treatment for steroid-resistant GvHD patients where no other such treatments are currently available.

DETAILED DESCRIPTION:
This is a prospective, phase II/III, randomized clinical study to compare the efficacy and safety of BEGEDINA® (Begelomab) versus "conventional treatment" for treating steroid-resistant acute graft versus host disease (GvHD). Despite prophylactic treatment, GvHD still develops in up to 30% of allogeneic hemopoietic stem cell transplant (HSCT) recipients. GvHD is a life-threatening and complex immunological disease that may be acute or chronic. Acute GvHD affects mainly the skin, liver and gastrointestinal (GI) tissues with long-term survival directly related to the severity of skin, liver and gut involvement. First line treatment for patients with acute GvHD (Grade II or higher) is the immunosuppressive corticosteroid methylprednisolone. Although effective in over 50% of patients, durable responses are observed in only a third of patients and it also confers a risk of severe infection. Steroid-resistant acute GvHD is associated with a high rate of morbidity and mortality, primarily from infections and/or multi-organ failure. Despite this, there are no authorized treatments for non-responders and GvHD remains largely an untreatable disease with limited survival and thus a great unmet therapeutic need. BEGEDINA® (Begelomab) is a murine immunoglobulin G (IgG) 2b monoclonal antibody against CD26 (dipeptidyl peptidase-4; DPP4) and is produced by biotechnological means and is a new potential therapeutic approach. BEGEDINA® has been shown to bind to CD26 which is present on a subset of CD4+ T helper lymphocytes leading to down-regulation of CD26 signaling and inhibition of immune response and thus therapeutic improvements. BEGEDINA has been investigated in two completed clinical studies: a pilot study and a dose-finding study and so far showing promising efficacy, safety and tolerability.

The primary objective for this study is therefore to determine the efficacy of BEGEDINA® versus conventional therapy in steroid-resistant acute GvHD. To satisfy this objective, two co primary hypothesis will be tested. The first is that the overall response rate consisting of the Complete Responders and the Partial Responders (CR+PR) at Study Day 28 will be higher in the BEGEDINA® treated subjects. The second is that the incidence of transplant-related mortality (TRM) at 6 months will be reduced in those subjects treated with BEGEDINA® versus those treated with conventional therapy. Additional secondary efficacy endpoints will also be assessed as a measure of effectiveness. In addition, some pharmacokinetics assessments will be performed. Adverse events (AEs) will be coded using MedDRA and the frequency, causality and intensity of AEs will be compared to conventional therapies. Further safety analysis will also include laboratory findings, vital signs, immunogenicity and other assessments. Finally, some exploratory analysis will also be performed.

This will be a prospective, multicenter, randomized, open-label, phase II/III clinical study in which subjects will be randomly assigned in a 1:1 ratio to receive BEGEDINA® treatment or the best conventional treatment available in their territory as no second line therapy is currently approved. It is planned to enroll 184 male or female adult subjects with an upper age limit of 65 years with steroid-resistant acute GvHD. BEGEDINA® will be administered at a dose of 2.7 mg/m2/day for 5 consecutive days from Study Day 1 through to Study Day 5, and on Study Days 10, 14, 17, 21, 24, and 28. Thus, the expected duration for each subject will be approximately 12 months. The final statistical analysis plan (SAP) will be finalized prior to database lock. Baseline characteristics of the subject sample will be described using summary statistics. All statistical tests will be conducted at a 2-sided significance level of 5% unless specifically specified. Multiple Imputation methods will be used as the primary method for accounting for missing data.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 and ≤65 years of age.
2. Recipient of an allogeneic hematopoietic stem cell transplantation (HSCT). Note: Subjects with GvHD following donor lymphocyte infusion post-HSCT are also eligible
3. Steroid-resistant acute GvHD, Grade II-IV, defined as: progressive disease (deterioration of at least 1 stage in 1 organ) after 3 days of primary treatment with methylprednisolone 2 mg/kg, or equivalent. or lack of at least a partial response (PR) after 7 days of primary treatment with methylprednisolone 2 mg/kg or equivalent. or lack of a complete response (CR) after 14 days of primary treatment with methylprednisolone 2 mg/kg or equivalent. Note: Subjects who may have received an increase in their steroid dose treatment prior to randomization will be eligible for enrollment. An increase in steroid dose will not be considered as second-line therapy.
4. Evidence of previous myeloid engraftment (absolute neutrophil count ≥0.5 x 10^9/L).
5. Karnofsky Performance Status Scale ≥50%.
6. Adequate renal function as defined by serum creatinine ≤2 × upper limit of normal or calculated creatinine clearance (CrCl) of ≥30 mL/min using the Cockroft-Gault equation: Calculated CrCl= ([140-age in years] x [ideal body mass {IBM} in kg])/72 x (serum creatinine value in mg/dL), where IBM = IBM (kg) = ([height in cm- 154] × 0.9) + (50 if male, 45.5 if female).
7. Subject must be willing and able to comply with study requirements, remain at the clinic, and return to the clinic for the follow-up evaluation, as specified in this protocol during the study period.
8. Able and willing to provide signed informed consent.

Exclusion Criteria:

Subjects will not be entered in the study for any of the following reasons:

1. Prior second-line systemic treatment for GvHD.
2. Received agents other than steroids for primary treatment of acute GvHD.
3. Stage 1-2 skin acute GvHD alone (with no other organ involvement).
4. Acute steroid resistant GvHD beyond 28 days from first-line therapy (primary treatment).
5. Evidence of severe hepatic veno-occlusive disease or sinusoidal obstruction.
6. Evidence of encephalopathy.
7. Life expectancy <3 weeks.
8. Presence of chronic GvHD
9. Second or subsequent allogeneic transplant.
10. Previous solid organ transplant (with the exception of a corneal transplant >3 months prior to screening).
11. Relapsed disease after last transplant.
12. Human immunodeficiency virus positive.
13. Evidence of lung disease that is likely to require more than 2 liter per minute of O2 via face mask or an estimated FiO2 of 28% via other delivery methods in order to sustain an O2 saturation of 92% within the next 3 days.
14. Any underlying or current medical or psychiatric condition that, in the opinion of the investigator, would interfere with the evaluation of the subject including uncontrolled infection, heart failure, pulmonary hypertension. Any other serious medical condition, as judged by the investigator, which places the subject at an unacceptable risk if he or she were to participate in the study or confounds the ability to interpret data from the study.
15. Administration of any other investigational agents (not approved by the United States Food and Drug Agency [FDA] or European Medicines Agency [EMA] for any indication) within 30 days of randomization. Participated in any interventional clinical trial for an acute GvHD therapeutic agent or for an immunomodulatory drug, within the past 30 days or within 5 half-lives of the study treatment, whichever is the greater. Participated or is currently participating in any bone marrow derived autologous and allogeneic stem cell or gene therapy study.
16. Known hypersensitivity to murine proteins.
17. Women who are pregnant, breastfeeding or at risk to become pregnant during study participation; female subjects of childbearing potential who have not been started on an anti-ovulatory regimen prior to initiation of chemo-inductive regimen must test negative for pregnancy (serum) at the time of enrollment.
18. Male and female subjects who do not agree to take adequate measures to avoid pregnancy prior to study entry and for the duration of participation in the study (or for at least 3 months following the last dose of study drug, whichever is longer) (acceptable methods of birth control are described in protocol Section 6.2.1.6).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-02; Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Bacigalupo, MD, Principal Investigator
Locations (27):
- United States (10):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - University of Kansas Cancer Center and Medical Pavilion, Westwood, Kansas
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Hackensack University Medical Center - John Theurer Cancer Center, Hackensack, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke Cancer Center, Durham, North Carolina
  - The Ohio State University, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Huntsman Cancer Center, University of Utah, Salt Lake City, Utah
- France (3):
  - Centre Hospitalier Universitaire de Grenoble, La Tronche
  - Hospital Saint-Louis APHP (Hôpitaux Universitaires Sant-Louis), Paris
  - Centre Hospitalier Lyon-Sud, Pierre-Bénite
- Universitätsklinikum Hamburg-Eppendorf, Hamburg, Germany
- Italy (7):
  - Ospedale Casa Sollievo della Sofferenza, IRCCS, San Giovanni Rotondo, Foggia
  - Policlinico S.Orsola Malpighi, AOU di Bologna, Bologna
  - L'IRCCS A.O.U. San Martino - IST, Genova
  - Ospedale San Raffaele, Milan
  - A.O. Universitaria Policlinico Tor Vergata, Roma
  - Policlinico Universitario Agostino Gemelli, Roma
  - Ospedale Molinette, Torino
- Spain (4):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Univeristario de Salamanca, Salamanca
  - Hospital Universitari Politecnic La Fe, Valencia
- Universitätsspital Basel, Basel, Basel-Stadt (de), Switzerland
- University Hospital Southampton NHS Foundation Trust, Southampton, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Out of the 29 sites selected (USA, France, Italy, Spain, Switzerland, UK, Germany) for participation in this study, 22 of them have activated screening and enrolment procedures, and 15 sites have effectively enrolled and randomized participants in the study. The first site approved was in Spain on 07 October 2015.
Pre-assignment Details: Out of 184 subjects planned, 37 subjects were screened and 36 subjects were randomized by IVRS in a 1:1 ratio. All subjects signed the informed consent and met all eligibility criteria except one case that had an incomplete screening procedure (some blood tests have not been performed for the screening visit as requested by the protocol).
Groups:
- BEGEDINA® (Begelomab): 18 subjects from a total of 37 screened subjects were enrolled on Begedina arm. All subjects signed the informed consent and met all eligibility criteria.
- Conventional Second-line Treatment: 18 subjects from a total of 37 subjects were screened on Conventional Treatment arm. All subjects signed the informed consent and met all eligibility criteria.
Period: Overall Study
Arm/Group | BEGEDINA® (Begelomab) | Conventional Second-line Treatment
Started | 18 | 18
Completed | 5 | 5
Not Completed | 13 | 13
Not completed — Lack of Efficacy | 6 | 3
Not completed — Death | 5 | 4
Not completed — Adverse Event | 2 | 1
Not completed — Other reasons | 0 | 5

BASELINE CHARACTERISTICS:
Groups:
- BEGEDINA® (Begelomab): Subjects have received BEGEDINA 2.7 mg/m2/day IV for 5 consecutive days (Study Days 1, 2, 3, 4, 5) and then on Study Days 10, 14, 17, 21, 24 and 28, for a total of 11 doses. A window (+/- 1 day) was permitted for doses from Day 10 to Day 28, however, all efforts have been made to plan these doses with at least 48 hours between doses.
  The total volume of BEGEDINA to be administered was diluted in 100 mL of sodium chloride 9 mg/mL (0.9%) solution for injection prior to administration. The infusion lasted for 60 minutes.
  Begelomab: BEGEDINA® (Begelomab) is a murine immunoglobulin G (IgG) 2b monoclonal antibody against CD26 (dipeptidyl peptidase-4; DPP4) and is produced by biotechnological means.
- Conventional Second-line Treatment: Subjects in the conventional treatment arm have received a second line treatment, which were chosen by each center, based on the clinical conditions of the individual subject and according to the standard practice at the study center. Currently no treatments for this life-threatening disease have been approved in either the USA or Europe. The recommendations of the American Society for Blood and Marrow Transplantation (ASBMT) confirm that no treatment for acute steroid-refractory GvHD can be considered gold standard in terms of TRM or survival as results remain unsatisfactory and this approach has been agreed by the FDA and the EMA.
  Treatments were generally biological products and could include anti-thymocyte globulin, monoclonal antibodies, such as anti-CD147, basiliximab, daclizumab and alemtuzumab; mycophenolate mofetil; anti-TNF-alpha; pentostatin; dinileukin diftitox; N-acetyl-cysteine; sirolimus; and visulizumab.
- Total: Total of all reporting groups
Arm/Group | BEGEDINA® (Begelomab) | Conventional Second-line Treatment | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.4 (9.06) | 43.5 (13.74) | 48.3 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 13 | 12 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 7
  Not Hispanic or Latino | 13 | 15 | 28
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 17 | 17 | 34
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 5 | 12
  Italy | 3 | 3 | 6
  France | 4 | 3 | 7
  Germany | 1 | 0 | 1
  Spain | 3 | 7 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Overall Response at 28 Days
Description: The change in grade from baseline to Study Day 28 (-1/+2 day) was used to determine the response of GvHD to treatment using the following classifications:
  * Complete response (CR): complete resolution of all signs of GvHD.
  * Partial response (PR): improvement of 1 overall grade (i.e., change from baseline in IBMTR to a less severe grading).
  * Stable disease (SD): No change in GvHD grading (i.e., no change from baseline in IBMTR grade).
  * Disease progression (PD): Deterioration in one overall grade in GvHD (i.e., worsening in IBMTR by at least 1 grade compared to baseline).
  * Death
Time Frame: 28 days for OR
Measure: Count of Participants; unit: Participants
Groups:
- Conventional Second-line Treatment: Conventional Second-line Treatment: There are no approved second-line treatments for aGvHD and due to the life-threatening nature of the disease it was agreed with the FDA and EMA that BEGEDINA® would be compared with "best conventional second-line treatments" which will be chosen by each center, based on the clinical conditions of the individual sub
Arm/Group | BEGEDINA® (Begelomab) | Conventional Second-line Treatment
Number analyzed (Participants) | 18 | 18
Participants
  Complete response | 3 | 5
  Stable Disease | 3 | 3
  Partial Response | 5 | 8
  Progressive disease | 1 | 1

2. Secondary Outcome: Number of Participants With Overall Survival (OS) up to 180 Days
Description: For this endpoint, no statistical confirmatory test could be performed due to insufficient sample size.
Time Frame: Time frame is up to 180 days
Measure: Count of Participants; unit: Participants
Arm/Group | BEGEDINA® (Begelomab) | Conventional Second-line Treatment
Number analyzed (Participants) | 18 | 18
Participants
  Deceased | 13 | 8
  Alive | 5 | 10

3. Secondary Outcome: BEGEDINA Serum Concentrations Pre- and 15 Minutes Post-Infusion
Description: The pharmacokinetic (PK) objective for this study was to characterize the serum concentrations of BEGEDINA in subjects with Grades II-IV acute GvHD who have failed to respond to steroid treatment. Data was analyzed before and 15 minutes after infusion.
Time Frame: Time frame is up to Day 28
Population: The PK report presents the available data for 13 subjects on Begedina arm.
Measure: Median (Full Range); unit: ng/ml
Arm/Group | BEGEDINA® (Begelomab)
Number analyzed (Participants) | 13
ng/ml
  Day 1 pre-infusion | 0.0 [0 to 155]
  Day 1 post-infusion | 138.6 [72 to 1371]
  Day 5 pre-infusion | 96.4 [46 to 1617]
  Day 5 post-infusion | 591.1 [240 to 6880]
  Day 10 pre-infusion | 6.9 [0 to 1356]
  Day 10 post-infusion | 289.6 [127 to 2080]
  Day 14 pre-infusion | 5.3 [0 to 184]
  Day 14 post-infusion | 240.7 [126 to 2154]
  Day 17 pre-infusion | 6.3 [0 to 129]
  Day 17 post-infusion | 340.6 [196 to 8739]
  Day 21 pre-infusion | 0.0 [0 to 130]
  Day 21 post-infusion | 271.4 [94 to 1073]
  Day 24 pre-infusion | 10.9 [0 to 135]
  Day 24 post-infusion | 316.0 [164 to 1398]
  Day 28 pre-infusion | 11.5 [0 to 33]
  Day 28 post-infusion | 357.0 [196 to 436]

4. Secondary Outcome: Number of Participants With Adverse Events
Description: The safety parameters were analysed at the end of the study period (Day 180).
Time Frame: The safety parameters were analysed at the end of the study period (Day 180)
Measure: Count of Participants; unit: Participants
Arm/Group | BEGEDINA® (Begelomab) | Conventional Second-line Treatment
Number analyzed (Participants) | 18 | 18
Participants
  Early discontinuation | 16 | 14
  Deaths | 13 | 8
  Non-serious AE | 18 | 18
  SAE | 16 | 13

5. Other Pre Specified Outcome: Exploratory Objectives
Description: The exploratory objectives for this study were:
  * To evaluate the change in quality of life (QoL) from baseline;
  * To evaluate duration of response;
  * To evaluate OR by standard-risk and high-risk GvHD at onset
Time Frame: Time frame is up to 180 days
Population: This analysis could not be performed because of the premature discontinuation of the study. No data are available
Arm/Group | BEGEDINA® (Begelomab) | Conventional Second-line Treatment
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: All adverse events were collected in a 6 months period (180 days).
Description: Information about all AEs, whether volunteered by the subjects, discovered by investigator questioning, or detected through physical examination, laboratory test or other means, were collected and recorded on the eCRF AE section.
Groups:
- BEGEDINA® (Begelomab): The most frequent adverse events recorded after administration of BEGEDINA® were platelet count decreased (19.4% cases), anemia (16.7% cases), leukocytes count decreased (11.1% cases). Cytomegalovirus infection was found in 16.7% cases and peripheral edema in 13.9% cases.There were recorded 25 serious adverse events. At the end of the study rate of serious adverse events which determined early discontinuation in BEGEDINA® group was 22.2 % ( 4 subjects). At the end of the study (approx. day 180), death occurred in 36.1 % (13 subjects) in BEGEDINA® group.
- Conventional Second-line Treatment: The most frequent adverse events recorded in the conventional treatment arm were peripheral edema(22.2% cases), pyrexia (19.4% cases). Cytomegalovirus infection was found in 13.9% cases.There were recorded 29 serious adverse events. At Day 28, death occurred in 11.1% cases in this treatment group. At the end of the study rate of serious adverse events which determined early discontinuation in conventional treatment arm was 5.6
  % (one subject). Mortality (approx. day 180) was 22.2 % (8 subjects) in the conventional treatment group.
Arm/Group | BEGEDINA® (Begelomab) | Conventional Second-line Treatment
All-Cause Mortality (participants affected / at risk) | 13/18 | 8/18
Serious Adverse Events (participants affected / at risk) | 16/18 | 13/18
Other Adverse Events (participants affected / at risk) | 18/18 | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BEGEDINA® (Begelomab) (N=18) | Conventional Second-line Treatment (N=18)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 1 (1)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Graft versus host disease (Immune system disorders) | 2 (2) | 1 (1)
Graft versus host disease in liver (Immune system disorders) | 0 (0) | 1 (1)
Acute graft versus host disease (Immune system disorders) | 2 (2) | 0 (0)
Acute graft versus host disease in skin (Immune system disorders) | 0 (0) | 1 (1)
Pyrexia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Obliterative bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pneumoperitoneum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 0 (0) | 2 (4)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (2)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 2 (2) | 1 (1)
Septic shock (Infections and infestations) | 3 (3) | 1 (1)
Cytomegalovirus enteritis (Infections and infestations) | 1 (1) | 1 (1)
Bacterial sepsis (Infections and infestations) | 1 (1) | 0 (0)
Phlebitis infective (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BEGEDINA® (Begelomab) (N=18) | Conventional Second-line Treatment (N=18)
Flushing (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 3 (3)
Hypotension (Vascular disorders) | 3 (3) | 4 (4)
Shock (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Superior vena cava occlusion (Vascular disorders) | 1 (1) | 0 (0)
Transurethral bladder resection (Surgical and medical procedures) | 0 (0) | 1 (1)
Hypogammaglobulinaemia (Immune system disorders) | 1 (1) | 1 (1)
Graft versus host disease in gastrointestinal tract (Immune system disorders) | 2 (2) | 0 (0)
Graft versus host disease in liver (Immune system disorders) | 2 (2) | 0 (0)
Acute graft versus host disease in skin (Immune system disorders) | 0 (0) | 1 (1)
Acute graft versus host disease (Immune system disorders) | 2 (2) | 1 (1)
Asthenia (General disorders) | 0 (0) | 2 (2)
Chest pain (General disorders) | 0 (0) | 1 (1)
Face oedema (General disorders) | 0 (0) | 2 (2)
Fatigue (General disorders) | 3 (4) | 3 (6)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
Hypothermia (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 5 (7) | 8 (9)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Localised oedema (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 3 (4) | 6 (7)
Adjustment disorder with depressed mood (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 4 (5) | 2 (3)
Apathy (Psychiatric disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 3 (4) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 2 (2) | 2 (2)
Disorientation (Psychiatric disorders) | 0 (0) | 1 (1)
Hallucination (Psychiatric disorders) | 1 (1) | 0 (0)
Hallucination auditory (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1)
Mental status change (Psychiatric disorders) | 0 (0) | 1 (1)
Bradyphrenia (Psychiatric disorders) | 0 (0) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Oedema genital (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Penile pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 4 (5)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (7) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (2)
Blood bilirubin increased (Investigations) | 5 (10) | 1 (1)
Blood creatine increased (Investigations) | 2 (2) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 1 (1)
Blood magnesium decreased (Investigations) | 1 (1) | 0 (0)
Blood potassium decreased (Investigations) | 1 (1) | 0 (0)
Blood tryglicerides increased (Investigations) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 2 (2) | 0 (0)
Haptoglobin decreased (Investigations) | 1 (1) | 0 (0)
International normalised ratio increased (Investigations) | 1 (3) | 0 (0)
Low density lipoprotein increased (Investigations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 3 (7) | 2 (5)
Neutrophil count decreased (Investigations) | 2 (5) | 2 (2)
Platelet count decreased (Investigations) | 7 (24) | 1 (6)
Weight decreased (Investigations) | 2 (2) | 0 (0)
Weight increased (Investigations) | 1 (1) | 1 (1)
White blood cell count decreased (Investigations) | 4 (8) | 2 (2)
Transaminases increased (Investigations) | 0 (0) | 2 (2)
Troponin increased (Investigations) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (2) | 0 (0)
Staphylococcus test positive (Investigations) | 0 (0) | 1 (2)
Klebsiella test positive (Investigations) | 0 (0) | 1 (1)
Liver function test increased (Investigations) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Left ventricular hypertrophy (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac disorder (Cardiac disorders) | 0 (0) | 1 (1)
Mitral valve disease (Cardiac disorders) | 0 (0) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary odema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 6 (11) | 4 (6)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 2 (3) | 2 (2)
Neutrophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (2) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1)
Intention tremor (Nervous system disorders) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1)
Palmar-plantar erythrodysaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 1 (1)
Spinal cord compression (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 3 (3)
Dry eye (Eye disorders) | 1 (1) | 2 (2)
Visual impairment (Eye disorders) | 0 (0) | 1 (2)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Eustachian tube disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Abdominal distention (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (5) | 4 (10)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric dilatation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 2 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal hameorrhage (Gastrointestinal disorders) | 0 (0) | 1 (4)
Vomiting (Gastrointestinal disorders) | 3 (3) | 2 (2)
Anal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Lower Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Oliguria (Renal and urinary disorders) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (2) | 2 (2)
Proteinuria (Renal and urinary disorders) | 2 (4) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 2 (2)
Urethral pain (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Bladder disorder (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 2 (2) | 3 (4)
Acute kidney injury (Renal and urinary disorders) | 4 (4) | 1 (1)
Hepatocellular injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatobiliary disease (Hepatobiliary disorders) | 1 (1) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Nail dystrophy (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3)
Skin atrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperparathyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Haemochromatosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 7 (11) | 3 (3)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 (6) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 (3) | 4 (5)
Hypocalcaemia (Metabolism and nutrition disorders) | 3 (3) | 2 (3)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2) | 3 (5)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (8) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Tetany (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Arthralgia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Back pain (Metabolism and nutrition disorders) | 1 (1) | 3 (6)
Bone pain (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Flank pain (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Muscular weakness (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Pain in extremity (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Sarcopenia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (13) | 3 (8)
Bacterial disease carrier (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 1 (1)
Enterococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Epstein-Barr virus infection (Infections and infestations) | 3 (3) | 1 (1)
Liver abscess (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 4 (4) | 2 (2)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Stenotrophomonas infection (Infections and infestations) | 1 (1) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 1 (1) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Parvovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Oesophageal infection (Infections and infestations) | 0 (0) | 1 (1)
Adenovirus infection (Infections and infestations) | 0 (0) | 1 (2)
Enterococcal infection (Infections and infestations) | 2 (2) | 0 (0)
Escherichia infection (Infections and infestations) | 1 (1) | 0 (0)
Candida infection (Infections and infestations) | 2 (2) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 6 (8) | 4 (6)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 3 (3)
Sepsis (Infections and infestations) | 1 (1) | 2 (2)
Bacterial sepsis (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 2 (2) | 3 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
This clinical study has prematurely ended, due to the lack of enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution and Investigators agree that any publication by Institution or Investigators of the Study Results shall not be made before the first multi-centre publication. In the event there is no multi-centre publication within twenty-four (24) months after a Study has been completed, Institution shall have the right to publish its results from the Study.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-13): https://cdn.clinicaltrials.gov/large-docs/84/NCT02411084/Prot_SAP_000.pdf